CLINICAL TRIAL: NCT04959552
Title: FreeStyle Libre 2 Flash Glucose Monitoring System Intervention Phase Study- FreeStyle Libre 2
Brief Title: FSL2 Post Approval Study for Pediatric and Young Adults Patients
Status: Recruiting | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-PMS-20196
Record Dates: First submitted 2021-06-14; First posted 2021-07-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre 2 — The FreeStyle Libre 2 Flash Glucose Monitoring

SUMMARY:
This is a prospective, multi-center, non-randomized, single-arm study intended to characterize the safety of the FreeStyle Libre 2 Flash Glucose Monitoring System when used to manage diabetes in pediatric and young adult patient populations.

DETAILED DESCRIPTION:
Approximately 550 pediatric and young adult subjects aged 4-30 years with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes will be enrolled in the study. Subjects and/or their caregivers will utilize he FreeStyle Libre 2 Flash Glucose Monitoring System for managing diabetes for 6 months. Subjects and/or their caregivers will maintain a diary/log book of Adverse Events experienced during the duration of the study. Assessment of Adverse Events will occur via self reporting at each monthly visit and/or phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 4 - 30 years of age.
2. Subject must have a diagnosis of type 1 or type 2 diabetes mellitus for at least 3 months prior to enrollment.
3. Subject is currently using Self Monitoring of Blood Glucose (SMBG) for managing their diabetes.
4. Subject has completed participation in clinical study ADC-US-PMS-20194 or has at least six (6) months of medical history hypoglycemia or hyperglycemia requiring healthcare professional intervention.
5. Subject and/or caregiver must be able to read and understand English.
6. In the investigator's opinion, the subject and/or caregiver must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
7. Subject and/or parent or guardian must be willing and able to provide written signed and dated informed consent and assent when appropriate.

   Exclusion Criteria:
8. Subject has previously used a continuous glucose monitoring system to manage their diabetes within the last six (6) months.
9. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
10. Subject is known to be pregnant or is attempting to become pregnant at the time of enrollment.
11. Subject is on dialysis at the time of enrollment.
12. Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff.
13. Subject currently is participating in another clinical trial.
14. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and young adult subjects aged 4-30 years with type 1 or type 2 diabetes, who require daily blood glucose monitoring to manage their diabetes. Approximately 35% of the study population will be age 4-12 years of age, and approximately 30% of the study population will be age 18-30 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety of the FreeStyle Libre 2 Flash Glucose Monitoring System when used to manage diabetes in pediatric and young adult patient populations | Six Months
  Incidence rate of severe hypoglycemic occurrences requiring health care professional (HCP) intervention including EMT assistance, hospital/clinic visit and/or hospitalization and moderate hypoglycemia in which the patient required the assistance of another person (e.g. as a result of confusion, coma, or seizure) during the study will be collected.
  The incidence rate of severe hypoglycemia associated with FSL2 use from this study will be compared with the incidence rate observed from self-monitoring blood glucose (SMBG) use observed during the prior 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (3):
- United States (3):
  - Yale Pediatric Endocrinology Clinic, New Haven, Connecticut
  - The Children's Mercy Hospital, Kansas City, Missouri
  - The DOCS, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided